CLINICAL TRIAL: NCT05173220
Title: Tracheal Intubation in Emergency Prehospital Setting. Impact of the Bougie on the Failure Rate of First Intubation Attempt.
Brief Title: Impact of the Bougie on the Prehospital Setting Intubation Quality.
Acronym: SMURIDS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bruno Simonnet (Unknown)
Responsible Party: Principal Investigator, Michel GALINSKI, M.D., Ph.D., University Hospital, Bordeaux
Other Study IDs: CHUBX-URG-02
Record Dates: First submitted 2021-12-08; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Tracheal Intubation Morbidity; Prehospital Emergency
Keywords: difficult intubation; prehospital emergency; risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tracheal intubation in an out-of-hospital setting is a frequent and potentially difficult procedure. The risk of adverse events increases dramatically with the number of attempts. The failure rate of the first intubation attempt ranges from 5 to 32% and the risk factors are unclear.

In recent study, the prevalence of a failed first intubation attempt was 31.4% [95% CI = 30.2-32.6] among 1546 patients managed in an out-of-hospital setting. In this multicenter study, our center (N=462) had a rate of 36% of failure of the first attempt. Seven variables were independently associated with a failed first intubation attempt. Some of the associated factors can be improved (operator training and experience), but most cannot. Moreover some of them can not be anticipated in this context. A randomized control trial performed in an emergency department and a prospective, observational, pre-post study design showed that systematic use of a bougie during the first intubation attempt improved the success rate.

Our objective is to measure the impact of a modification of our intubation modalities introducing the incitation of the use of the bougie on the first intubation attempt in the prehospital setting.

DETAILED DESCRIPTION:
Tracheal intubation (TI) is a procedure that is frequently performed in an out-of-hospital emergency setting. TI is associated with a risk of adverse events, including severe sequelae such as hypoxemia, vomiting, aspiration, hypotension, and cardiac arrest. The risk of adverse events increases dramatically with the number of intubation attempts. Thus, it is important that the first intubation attempt succeeds. In most cases, the environment in an out-of-hospital setting is not appropriate for intubation, and can be austere (outside, restricted space, patient on the floor, or public place) or dangerous (mountain, sea, or roadside). Although literature data are abundant, they are extremely heterogenous. Indeed, the available studies differ in terms of operator profiles, TI indications, and design. Based on studies involving management by physician-led teams in out-of-hospital settings and for which data are available, the failure rate of the first intubation attempt ranges from 5% to 32%. Numerous variables are associated with difficult intubation (DI), such as more than two attempts and bad glottic visualization, but few studies have analyzed risk factors for failure of the first attempt. Identification of such factors would decrease the risk of complications.In recent study, the prevalence of a failed first intubation attempt was 31.4% [95% CI = 30.2-32.6] among 1546 patients managed in an out-of-hospital setting. In this multicenter study, our center (N=462) had a rate of 36% of failure of the first attempt. Seven variables were independently associated with a failed first intubation attempt, operator with ≤ 50 prior intubations, small inter-incisor space, limited head extension, macroglossia, ENT tumor, cardiac arrest, and vomiting.

Some of the associated factors can be improved (operator training and experience), but most cannot. Moreover some of them can not be anticipated in this context. A randomized control trial performed in an emergency department showed that systematic use of a bougie during the first intubation attempt improved the success rate. A prospective, observational, pre-post study design including 823 and 771 patients respectively, showed that the use of a bougie on the first intubation attempt by paramedic in prehospital setting, improved the success rate. So we modified our intubation modalities introducing the incitation of the use of the bougie on the first intubation attempt in the prehospital setting.

The main objective of this study is to compare the rate of first intubation attempt in a new observational study performed in our center with the rate of the first assessment and to measure the impact of the introduction a systematic bougie in our intubation modalities. The secondary objective is to measure in this new cohorte rate of first intubation attempt between intubation with and without bougie.

The follow up will be restricted to the area of prehospital emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* all patients intubated by Emergency Medical System (EMS) team

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with life-threatening distress requiring emergency intubation.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
Failure of the first intubation attempt | 1 hour
  Yes/No

SECONDARY OUTCOMES:
Number of prior intubations done by operator ≤ 50 | 1 hour
  yes/No
Operator position during intubation | 1 hour
  Upright/on knees/Lying on the floor/Lateral left decubitus/other
Gender | 1 hour
  Male/female
Age | 1 hour
  Year
Body mass index | 1 hour
  kg.m 2
Macroglossia | 1 hour
  yes/no
ENT tumor | 1 hour
  Yes/no
Inter-incisor space less than 2 fingerbreadths | 1 hour
  yes/no
limited head extension | 1 hour
  Yes/no
possible mandibular subluxation | 1 hour
  yes/no
thyromental length less than 3 fingerbreadths | 1 hour
  yes/no
Large neck size | 1 hour
  Yes/no
Foreign body in upper airway | 1 hour
  Yes/no
Upper airway bleeding/fluid | 1 hour
  Yes/no
Facial trauma | 1 hour
  Yes/no
Vomiting | 1 hour
  Yes/no
cardiorespiratory arrest | 1 hour
  yes/no
Patient on the floor | 1 hour
  Yes/no
Place where the intubation was done | 1 hour
  outside/at home/others/ambulance
restricted space | 1 hour
  Yes/no
if cardiac arrest, thoracic compression during intubation | 1 hour
  Yes/no
side events /complications during the intubation until 30 minutes after | 1 hour
  Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL GALINSKI, M.D, Ph.D, Principal Investigator — University Hospital, Bordeaux; BRUNO SIMONNET, M.D, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de BORDEAUX - Hôpital Pellegrin - Pôle Urgences adultes - SAMU, Bordeaux, France